CLINICAL TRIAL: NCT07327424
Title: Feasibility of Suprapubic Transvesical Endoscopic Prostatectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed M Abdelbary, MD, Ahmed Abdelbary, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/01072025/Mohamed
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Prostate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suprapubic Transvesical endoscopic prostatectomy (Experimental)
  Interventions: Other: Suprapubic transvesical endoscopic prostatectomy

INTERVENTIONS:
Other: Suprapubic transvesical endoscopic prostatectomy — Cysto-uretheroscopy will be done to evaluate the urethera , detect any bladder pathology and to visualise steps of insertion of laparoscopic port. The patient will be in supine position, and the surgeon will stand beside the patient .The bladder is filled with normal saline until it is completely full . Using Ultrasound A 18 G puncture needle is inserted 4 cm above the upper margin of the symphysis pubis to gain access to the bladder. then track is formed through single step dilation using a 30 Fr amplatz dilator and 10 mm laparoscopic port over it. Before starting the procedure, the ureteral orifices must be identified.

SUMMARY:
In patients with penile prosthesis, any transurethral procedure could place the implant at risk. The use of long or extra-long resectoscope can be of some assistance; however, these are not available in many institutions. So suprapubic transvesical endoscopic prostatectomy is newly developed to bypass the anterior urethra. Thus, the aim of this study is to determine safety and efficacy of Suprapubic Transvesical endoscopic prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with moderate to severe lower urinary tract symptoms ( IPSS score ≥ 8 ) indicated for surgical intervention with prostate size less than 120 cc.

Exclusion Criteria:

* History of previous pelvic surgery, urothelial cancer, kidney transplantation, uncontrolled coagulopathy, and significant central fat accumulation that could potentially increase the risk during transvesical access(body mass index not exceeding 27 kg/m2)

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score | 6 months

SECONDARY OUTCOMES:
Q max | 6 months
PVR (post-void residual volume) | 6 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT07327424/Prot_SAP_000.pdf